CLINICAL TRIAL: NCT06122324
Title: Evaluation of the Effect of Lidocaine on Hemodynamic Response and Postoperative Sore Throat
Brief Title: Effect of Lidocaine on Hemodynamic Response and Postoperative Sore Throat
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, kübra taşkın, specialist medical doctor anesthesiology and reanimation, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: kartalanesthesia
Record Dates: First submitted 2023-11-01; First posted 2023-11-08 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Sore Throat
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lidocaine group: Patients in Group 1 will receive 40 mg of lidocaine HCl solution 5 minutes before endotracheal intubation.
  Interventions: Drug: Lidocaine Hydrochloride
- control group: The second group will receive standard anesthesia management as the control group.

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — Patients in Group 1 will receive 40 mg of lidocaine HCl solution 5 minutes before endotracheal intubation.
  Groups: lidocaine group

SUMMARY:
Postoperative sore throat (POST) is a common outcome of general anesthesia in patients who undergo endotracheal intubation, and the estimated risk varies between 14.4% and 62%. It is one of the most undesirable postoperative anesthesia complications and has a negative impact on patient satisfaction and quality. Mucosal damage, inflammation, and erosion caused by endotracheal intubation all contribute to the development of POST. Therefore, POST is a condition that requires prevention and improvement.

In the study, patients will be divided into two groups. The investigators will include 100 patients undergoing surgery under general anesthesia. The first group will receive 40 mg of lidocaine HCl solution 5 minutes before endotracheal intubation, while the second group will receive standard anesthesia management as the control group.

Throat pain assessment will be conducted in patients at 2, 6, 12, and 24 hours after surgery.

DETAILED DESCRIPTION:
Between November 2023 and December 2023, a total of 100 patients aged 18-65 with ASA 1-3 classification who are electively scheduled for laparoscopic cholecystectomy will participate in the study. Patients with ASA 4 or higher, those aged 65 and older, those under 18, and individuals with a known allergy to local anesthesia will not be included in the study. Patients who require intubation and are admitted to the intensive care unit or who experience mortality will be excluded from the study.

All patients will undergo preoperative assessment one day before the surgery, and written informed consent will be obtained for participation in the study. Patients will be randomly assigned to groups using a computer-generated randomization table. Patients in Group 1 will receive 40 mg of lidocaine HCl solution 5 minutes before endotracheal intubation, while the second group will receive standard anesthesia management as the control group.

Demographic data, medical history, American Society of Anesthesiologists (ASA) classification, and pre- and post-lidocaine administration cardiac output (CO) and oxygen consumption (VO2), anesthesia time, surgical duration, as well as the occurrence of postoperative hypotension (systolic blood pressure decreased by more than 20% from baseline or SBP < 80 mmHg during surgery), nausea and vomiting, hypoxemia (SpO2 < 90% or PaO2 < 60 mmHg), hypercapnia (PaCO2 > 45 mmHg), and agitation during the awakening period will be recorded.

Throat pain will be assessed and recorded at postoperative hours 2, 6, 12, and 24. Throat pain will be evaluated using a throat pain scoring system ranging from 0 (no pain) to 3 (worst imaginable pain). After the surgery, all patients will be transferred to the post-anesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* electively laparoscopic cholecystectomy.

  * ASA I-III,
  * between 18-65 years

Exclusion Criteria:

* ASA IV and above

  • over 65 - under 18 years of age
* lidocaine allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 100 patients aged 18-65 with ASA 1-3 classification will participate in the study, undergoing elective laparoscopic cholecystectomy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The effect of lidocaine on postoperative sore throat | postoperative 24 hours
  The primary outcome of the study is to demonstrate whether lidocaine reduces postoperative sore throat. Sore throat and hoarseness of the patients were also investigated and recorded at the postoperative 0th, 2nd, 4th, and 24th hours. Sore throat was assessed with a scale as 0: no sore throat; 1: minimal sore throat (complaints of sore throat only on question); 2: moderate sore throat (accompanying sore throat); and 3: severe sore throat (voice change or hoarseness related to sore throat).

SECONDARY OUTCOMES:
Effect of lidocaine on hemodynamic response | perioperative
  The secondary outcome of the study is to assess the impact of lidocaine on hemodynamic response. Before induction, after induction, after intubation at 1st and 5th minutes, and postoperative heart rate increase and blood pressure increase will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: hülya yılmaz ak, Principal Investigator — Kartal Dr Lutfi Kırdar City Hospital
Locations (1):
- University of Health Science, Kartal Dr Lütfi Kırdar Training and Research Hospital, Kadiköy, İ̇stanbul, Turkey (Türkiye)